CLINICAL TRIAL: NCT00189644
Title: 6 FEC 100 Vs 4 FEC 100 Followed by 4 Taxol in N+ Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association Européenne de Recherche en Oncologie (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AERO-B2000
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: 6 FEC 100
Procedure: 4 FEC 100 followed by 4 Taxol

SUMMARY:
The main objective of this randomized trial is to compare 6 FEC100 to 4 FEC100 + 4 Taxol in patients with resected node positive breast cancer. Main endpoint is disease free survival. Secondary endpoints are overall survival, time to local recurrence, time to distant metastases, and tolerance. A total of 840 patients have been included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer of the breast,
* Mastectomy or complete tumorectomy,
* Histologically proven homolateral, axillary lymph node involvement (at least 1 N+)
* Period between surgery (second operation in case of primarily incomplete resection) and the start of chemotherapy < 2 months,
* Biological criteria (before the first FEC cycle):

  * Neutrophils >1.5 109 /L
  * Platelets >100 109/L
  * Hemoglobin >10 g/dl
  * Creatininemia <120 mmol/1
  * Bilirubinemia <1.5 Upper normal value
* Female patients over 18 years old
* Written and signed informed consent
* Performance Status less than or equal to 2 (WHO scale, see Annex IV)

Exclusion Criteria:

* Prior chemotherapy or radiotherapy, including neo-adjuvant treatment for cancer of the breast,
* Bilateral breast cancer or history of contralateral breast cancer
* Cardiac history: cardiac insufficiency (LVEF <50%) or coronary decompensation
* Pregnancy and breast-feeding (effective contraception is mandatory in the case of women of child-bearing potential)
* Inflammatory breast cancer
* Distant metastasis or supraclavicular adenopathy
* Benign pathology or history of malignant pathology accompanied by a life expectancy of less than two years
* Contra-indication to Anthracyclines, Cyclophosphamide, 5FU or Taxol
* Psychiatric pathology
* Patient participating in another trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Piedbois, MD, Principal Investigator — Association Europeenne de Recherche en Oncologie; Anne-Chantal Braud, MD, Principal Investigator — Association Europeenne de Recherche en Oncologie; Daniel Serin, MD, Principal Investigator — Association Europeenne de Recherche en Oncologie